CLINICAL TRIAL: NCT06898996
Title: FITting Non-invasive Testing Into Lynch Syndrome Colorectal Cancer Surveillance: a Multi-center, Prospective Study
Brief Title: FITting Non-invasive Tests in Lynch Syndrome Surveillance
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Columbia University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-1133; R01CA287257-01 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Lynch Syndrome; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, and stool samples will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-invasive surveillance test: Easily accessible, affordable and acceptable tests can be used to triage Lynch syndrome patients to colonoscopy
  Interventions: Other: Fecal immunochemical test

INTERVENTIONS:
Other: Fecal immunochemical test — Detects blood in stool

SUMMARY:
The purpose of this clinical study is to evaluate the accuracy of the fecal immunochemical test (FIT) in comparison to colonoscopy in patients with Lynch Syndrome (LS) who are undergoing colonoscopy surveillance.

DETAILED DESCRIPTION:
Lynch syndrome (LS), the most common inherited cause of colorectal cancer (CRC) affecting about 1.2 million Americans. Colonoscopy starting early in adulthood and repeated yearly or biennially is the only recommended surveillance strategy which translates into about 25-50 lifetime colonoscopies. This intensive colonoscopy surveillance is not ideal because CRC risk varies widely by LS gene and age, colonoscopies are invasive, costly, and not readily accessible to all patients, and adherence is suboptimal.

This clinical study will examine the performance of the fecal immunochemical test (FIT) in Lynch Syndrome (LS) patients undergoing colonoscopy surveillance. In addition to assessing the characteristics of the FIT test, such as specificity, sensitivity, and both negative and positive predictive values, the study will also explore LS patients' attitudes toward and acceptability of non-invasive testing methods. This comprehensive approach aims to provide insights into both the diagnostic effectiveness of FIT and the potential for improving patient adherence to screening protocols through less invasive options.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of LS with a confirmed pathogenic variant in MLH1, MSH2, MSH6, PMS2 or EPCAM genes.
* Aged 20 - 75 years (for those with pathogenic variants in MLH1, MSH2, and EPCAM)
* Aged 30 - 75 years (for those with pathogenic variants in PMS2 or MSH6).
* Have an upcoming standard of care (SOC) colonoscopy appointment in line with standard LS surveillance guidelines (NCCN).
* Willing to sign informed consent, collect stools samples and complete surveys

Exclusion Criteria:

* Individuals who have not proceeded with genetic testing and therefore are not known to have LS, despite family history and/or criteria for testing.
* Individuals who have previously undergone a subtotal or total colectomy.
* Newly diagnosed Lynch Syndrome patients < 20 years old with a pathogenic variant in MLH1, MSH2 or EPCAM, MSH6 or PMS2.
* Newly diagnosed Lynch Syndrome patients < 30 years old with a pathogenic variant in MSH6 or PMS2.
* Individuals who are pregnant.
* Individuals with inflammatory bowel disease or active malignancy.
* Individuals not willing or able to sign informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged 20 - 75 years who have been diagnosed with Lynch syndrome
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Measure of specificity | baseline -12 months
  Measure specificity of Fecal immunochemical test (FIT) in Lynch Syndrome (LS) patients undergoing colonoscopy surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Kupfer, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No